CLINICAL TRIAL: NCT06885255
Title: Effects of Intermittent Fasting and Its Combination with High-Intensity Interval Training on Inflammatory and Metabolic Markers, As Well As the Microbiome in Patients with Metabolic Syndrome: a Randomized Controlled Pilot Study
Brief Title: Effects of Intermittent Fasting and Exercise on Inflammation, Metabolism, and the Microbiome in Metabolic Syndrome
Acronym: FIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, yurdagül zopf, Professor of Integrative Medicine with a Focus on Nutritional Medicine (W3), Director of the Hector Center for Nutrition, Exercise, and Sports, University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-60_2-B
Record Dates: First submitted 2025-03-06; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Syndrome; Obesity and Obesity-related Medical Conditions
Keywords: obesity; metabolic syndrome; high-intensity interval training; inflammation; intermittent fasting
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Inflammation; Intermittent Fasting | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Metabolic syndrome - alternate day fasting (Experimental): Patients with metabolic syndrome who undergo alternate-day fasting in addition to regular advice on the mediterranean diet
  Interventions: Other: Alternate day fasting
- Metabolic syndrome - time restricted eating (Experimental): Patients with metabolic syndrome who undergo time restricted eating in addition to regular advice on the mediterranean diet
  Interventions: Other: Time restricted eating
- Metabolic syndrome - time restricted eating plus high-intensity interval training (Experimental): Patients with metabolic syndrome who undergo time restricted eating plus high-intensity interval training in addition to regular advice on the mediterranean diet
  Interventions: Other: Time restricted eating; Other: High-intensity interval training
- Metabolic syndrome - controls (No Intervention): Patients with metabolic syndrome exclusively receiving regular advice on the mediterranean diet
- Healthy - controls (No Intervention): Healthy controls exclusively receiving regular advice on the mediterranean diet

INTERVENTIONS:
Other: Alternate day fasting — Participants are instructed to alternate between consuming 100% of their usual energy intake on one day and only 25% on the following day.
  Arms: Metabolic syndrome - alternate day fasting
Other: Time restricted eating — Subjects are instructed to limit their energy intake to 8 hours a day and to fast for the remaining 16 hours.
  Arms: Metabolic syndrome - time restricted eating; Metabolic syndrome - time restricted eating plus high-intensity interval training
Other: High-intensity interval training — Patients participate in high-intensity interval training.
  Arms: Metabolic syndrome - time restricted eating plus high-intensity interval training

SUMMARY:
The goal of this intervention trial is to assess the effects of intermittent fasting, both alone and in combination with high-intensity interval training, on patients with obesity and metabolic syndrome. The main question it aims to answer is:

Does intermittent fasting, with or without high-intensity interval training, reduce chronic inflammation in patients with obesity and metabolic syndrome?

Participants will follow an intermittent fasting regime for 3 months, with one intervention group additionally participating in high-intensity interval training twice a week. In addition, there are two control groups: one consisting of participants with metabolic syndrome and one consisting of generally healthy individuals. The study includes a 3-month intervention phase followed by a 3-month follow-up phase. During the 6-month study period, all participants will attend 6 in-house study visits and 2 phone visits, during which they will undergo assessments and receive nutritional counseling.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study.
* Persons aged 18 years and older.
* Diagnosis of Metabolic Syndrome (MetS) with elevated hsCRP.

Exclusion Criteria:

* Pregnant or nursing individuals.
* Cardiovascular diseases or orthopedic restrictions that prevent exercise.
* Use of medication or supplements that significantly affect study outcomes (e.g., anti-inflammatory medications, antibiotics within the last 6 weeks).
* Body weight greater than 200 kg (maximum capacity of training equipment).
* Individuals with mental illnesses that may impair their ability to understand or participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
hsCRP | From enrollment to the end of intervention at 3 months.
  High sensitivity C-reactive protein in mg/l.

SECONDARY OUTCOMES:
inflammatory markers and metabolic markers | From enrollment to the end of intervention at 3 months.
  Determination of inflammatory markers and metabolic markers in blood (e.g., sICAM-1, IGF-1, β-hydroxybutyrate, estrogens, androgens).
waist circumference | From enrollment to the end of intervention at 3 months.
  Measurement of waist circumference in centimeters (cm).
fasting blood glucose | From enrollment to the end of intervention at 3 months.
  Measurement of fasting blood glucose in milligrams per deciliter (mg/dL).
triglycerides | From enrollment to the end of intervention at 3 months.
  Measurement of triglycerides in milligrams per deciliter (mg/dL).
cholesterol | From enrollment to the end of intervention at 3 months.
  Measurement of cholesterol (total, LDL, HDL) in milligrams per deciliter (mg/dL).
blood pressure | From enrollment to the end of intervention at 3 months.
  Measurement of systolic and diastolic blood pressure in millimeters of mercury (mmHg).
cardiometabolic risk profile | From enrollment to the end of intervention at 3 months.
  Calculation of the MetS z-score by combining waist circumference, fasting blood glucose, triglycerides, cholesterol, and blood pressure. The z-score will be reported as a single value based on these separate measures.
maximal oxygen uptake | From enrollment to the end of intervention at 3 months.
  Measurement of maximal oxygen uptake (VO2max) via spiroergometry.
liver fat status | From enrollment to the end of intervention at 3 months.
  Measurement of liver fat status via ultrasound examination.
composition of the intestinal and oral microbiome | From enrollment to the end of intervention at 3 months.
  Determination of the composition of the intestinal and oral microbiome by sequencing bacterial 16sRNA on the MiSeq platform, as well as analysis of the stool metabolome.
skin microbiome | From enrollment to the end of intervention at 3 months.
  Determination of the composition of the skin microbiome.
cortisol | From enrollment to the end of intervention at 3 months.
  Detection of cortisol from 24-hour urine collection.
body weight | From enrollment to the end of intervention at 3 months.
  Measurement of body weight in kilograms (kg) using bioimpedance analysis.
body fat percentage | From enrollment to the end of intervention at 3 months.
  Measurement of body fat percentage (%) using bioimpedance analysis.
fat-free mass | From enrollment to the end of intervention at 3 months.
  Measurement of fat-free mass (in kilograms) using bioimpedance analysis.
muscle mass | From enrollment to the end of intervention at 3 months.
  Measurement of muscle mass (in kilograms) using bioimpedance analysis.
phase angle | From enrollment to the end of intervention at 3 months.
  Measurement of phase angle (in degrees) using bioimpedance analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hector-Center for Nutrition, Exercise and Sports, University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No